CLINICAL TRIAL: NCT05604040
Title: Home BP Monitoring with Lifestyle Changes and Mindfulness Practices to Improve Hypertension Control
Brief Title: Home Blood Pressure Monitoring to Improve Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Cleveland State University (Other); MetroHealth System, Ohio (Other)
Responsible Party: Principal Investigator, Irina Todorov, MD, Medical Director, Department of Wellness and Preventative Medicine, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 00169
Record Dates: First submitted 2022-10-09; First posted 2022-11-03 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-09

CONDITIONS: Hypertension
Keywords: blood pressure monitoring, home; shared medical appointments; lifestyle changes; coping skills
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Self-monitoring and education program for lifestyle changes (Experimental): Participants will send self-reports of their home BPs, diet, physical activity and emotions while attending a 6-week education program of lifestyle changes and coping skills. Participants will get summary reports of their home BP and lifestyle monitoring. Participants primary care physicians will be notified of persisting high BPs and final average home BP levels. Researchers will monitor home BP levels and change in hypertension control state
  Interventions: Behavioral: Lifestyle Modifications

INTERVENTIONS:
Behavioral: Lifestyle Modifications — Home BP monitoring with self-monitoring of emotions, diet, physical activity, with shared medical appointment program for lifestyle changes and coping skills

SUMMARY:
The goal of this single group pre-post-study is to test the possibility of self-monitoring with shared medical appointments program for lifestyle education in improving blood pressure (BP) of patients with uncontrolled hypertension.

The main questions it aims to address is:

1. To assess if patients with uncontrolled hypertension and their physicians will be interested in trying a program that includes self-monitoring with 6-week support for lifestyle changes and coping skills to improve BP and hypertension control.
2. To assess if patients with uncontrolled hypertension can safely participate in a program that includes self-monitoring with 6-week support for lifestyle changes and coping skills to improve their BP and ability to self-manage hypertension

Participants will:

* Send self-reports of their home BPs, diet, physical activity and emotions
* Attend 6-week education program of lifestyle changes and coping skills delivered by physicians, holistic psychotherapists and yoga therapists.

DETAILED DESCRIPTION:
Participants will be taught the proper use of Home BP machines using a teach-back technique. Patients will be loaned valid home BP machines.

Participants will be taught how to send self-reports of their home BP, diet, physical activity and emotions using an app on their phone.

Participants will be signed up for a 6-week educational program of lifestyle changes and coping skills delivered by physicians, holistic psychotherapists and yoga therapists.

Participants will receive summary reports of their Home BP, lifestyle and emotions.

Researchers will monitor home BP levels and any adverse effects. Primary care physicians of the patients with persisting high BP levels will be notified of their average home BPs. Patients will complete surveys that assess their ability to self-manage their hypertension, emotions, and social connections. Change in average home BP from before, during, and after 6-week educational program participation will be evaluated. Final average home BP and clinic BP notifications will be sent to the primary care physicians of all patients.

ELIGIBILITY:
Inclusion Criteria:

* Uncontrolled hypertension based on Clinic BP measurement of systolic BP>140 or diastolic BP >90 mm Hg (as the cutoff in the current common hypertension performance measures and ACO metrics)
* PCP recommends or patient desires a trial of self-monitoring and lifestyle modifications
* Patient owns a smart phone and be willing to complete self-reports of BP during study participation.

Exclusion Criteria:

* On dialysis
* Pregnant
* Have a terminal illness,
* Clinic BP > systolic>180, diastolic>110
* Arm circumference that exceeds the limit for the largest home BP monitor cuff
* Severe cognitive impairment
* Major cardiovascular or cerebrovascular event in the past 6 months (Coronary artery disease, heart valve problems, arrhythmias, heart failure, stroke)
* Any physical or mental impairment that would affect patients' ability to participate(Ability to participate will be assessed by demonstrated ability to use available home BP machine and complete self-report during recruitment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-10-14 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2024-06-16 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with uncontrolled hypertension referred or self-referred for self-monitoring and lifestyle education program by physicians or patient self-referrals | Up to 10 months
  Investigators will measure the percentage of patients with uncontrolled hypertension that were referred or self-referred to and enrolled per month in the program for self-monitoring and lifestyle changes.

SECONDARY OUTCOMES:
Change in mean BP measured by mm of Hg | Up to 12 weeks
  Change in average home BP in mm Hg from before, during, and after the 6-week educational program participation will be evaluated.
Percentage of study participants that change from uncontrolled hypertension state to controlled hypertension state. | Upto 12 weeks
  Change in the percentage of study participants with uncontrolled hypertension from before, during, and after the 6-week educational program participation will be evaluated.
Percentage of study participants that adhere to the self-monitoring and lifestyle education program | Up to 10 months
  Investigators will measure percentage of enrolled patients with uncontrolled hypertension that:
  * participated in at least 4 of the 6 weeks of education program
  * Preferred weekly educational materials instead of attending weekly shared medical appointments.
  * Sent self-reports of home BP at least 3days/week in 4 out of 6weeks
Percentage of study participants that did not benefit from self-monitoring and lifestyle education program as measured by persisting high BP of more than 160/100 and need for additional medications | Up to 10 months
  Investigators will measure percentage of enrolled patients with uncontrolled hypertension that:
  * had persisting average home BP>160/100
  * needed additional medications
Change in mean Self-efficacy scale | Up to 6 months
  The PROMIS Self-Efficacy for Managing Chronic Conditions item banks are well-validated and comprise of five domains, Self-Efficacy for Managing: Daily Activities, Symptoms, Medications and Treatments, Emotions, and Social Interactions. We will measure before, after the 6-week educational program participation, and 6 months later will be evaluated.

OTHER OUTCOMES:
Change in mean Mindfulness Attention Awareness Scale | Upto 6 months
  Investigators will assess exploratory outcomes of changes in coping skills using Mindfulness Attention Awareness Scale; Insomnia severity Index scale; Change in number of vegetable and fruit serving intake; Change in the number of minutes of physical activity; Number of hypertension medications; Comparison of BP trends from 12 months before to 12 months after participating in the self-monitoring and education program
Change in mean insomnia severity index scale | Upto 6 months
  Investigators will assess exploratory outcomes of changes in sleep using Insomnia severity Index scale;
Change in the mean number of vegetable and fruit serving intake | Upto 6 months
  Investigators will assess exploratory outcomes of Change in number of vegetable and fruit serving intake;
Change in the mean number of minutes of physical activity per week | Upto 6 months
  Investigators will assess exploratory outcomes of Change in the number of minutes of physical activity;
Change in the mean number of hypertension medications | Upto 12 months
  Investigators will assess exploratory outcomes of change in Number of hypertension medications; Comparison of BP trends from 12 months before to 12 months after participating in the self-monitoring and education program
Change in the mean BP from 12 months before to 12 months after program participation. | Upto 12 months
  Investigators will assess exploratory outcomes of change in Comparison of BP trends from 12 months before to 12 months after participating in the self-monitoring and education program
Patient and physician feedback on intervention | Upto 3 months
  Investigators will gain insights into what worked what did not work for patients and referring primary care physicians

CONTACTS AND LOCATIONS:
Overall Officials: Sonal J Patil, MD, MSPH, Principal Investigator — The Cleveland Clinic; Irina Todorov, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Beachwood, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muntner P, Hardy ST, Fine LJ, Jaeger BC, Wozniak G, Levitan EB, Colantonio LD. Trends in Blood Pressure Control Among US Adults With Hypertension, 1999-2000 to 2017-2018. JAMA. 2020 Sep 22;324(12):1190-1200. doi: 10.1001/jama.2020.14545. PMID 32902588
- [Background] Muntner P, Hardy ST. Together, We've Got This: The US Surgeon General's Call-to-Action on Hypertension Control. Am J Hypertens. 2021 Sep 22;34(9):893-894. doi: 10.1093/ajh/hpaa172. No abstract available. PMID 34313678
- [Background] Patil SJ, Wareg NK, Hodges KL, Smith JB, Kaiser MS, LeFevre ML. Home Blood Pressure Monitoring in Cases of Clinical Uncertainty to Differentiate Appropriate Inaction From Therapeutic Inertia. Ann Fam Med. 2020 Jan;18(1):50-58. doi: 10.1370/afm.2491. PMID 31937533
- [Background] Patil S, Bhayani, V., Yoshida,Y., LA; Wilson, G., Stange, KC., Saper, R. A RE-AIM Evaluation of Lay Advisor Interventions to Improve Hypertension Outcomes - A Systematic Review. presented at: American Heart Association Annual (AHA) Scientific Sessions 2021; 2021; Session QCOR at Sessions: Quality of Care and Outcomes Research.
- [Background] Liaw WR, Jetty A, Petterson SM, Peterson LE, Bazemore AW. Solo and Small Practices: A Vital, Diverse Part of Primary Care. Ann Fam Med. 2016 Jan-Feb;14(1):8-15. doi: 10.1370/afm.1839. PMID 26755778
- [Background] Tajeu GS, Tsipas S, Rakotz M, Wozniak G. Cost-Effectiveness of Recommendations From the Surgeon General's Call-to-Action to Control Hypertension. Am J Hypertens. 2022 Mar 8;35(3):225-231. doi: 10.1093/ajh/hpab162. PMID 34661634
- [Background] Nguyen-Huynh MN, Young JD, Ovbiagele B, Alexander JG, Alexeeff S, Lee C, Blick N, Caan BJ, Go AS, Sidney S. Effect of Lifestyle Coaching or Enhanced Pharmacotherapy on Blood Pressure Control Among Black Adults With Persistent Uncontrolled Hypertension: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2022 May 2;5(5):e2212397. doi: 10.1001/jamanetworkopen.2022.12397. PMID 35583869
- [Background] James PA, Oparil S, Carter BL, Cushman WC, Dennison-Himmelfarb C, Handler J, Lackland DT, LeFevre ML, MacKenzie TD, Ogedegbe O, Smith SC Jr, Svetkey LP, Taler SJ, Townsend RR, Wright JT Jr, Narva AS, Ortiz E. 2014 evidence-based guideline for the management of high blood pressure in adults: report from the panel members appointed to the Eighth Joint National Committee (JNC 8). JAMA. 2014 Feb 5;311(5):507-20. doi: 10.1001/jama.2013.284427. PMID 24352797